CLINICAL TRIAL: NCT05476133
Title: Application of a Training Program for Executive Functions in a Sample of Egyptian Children With Learning Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Engy Elhakeem, lecturer of phoniatrics, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0106137
Record Dates: First submitted 2022-07-15; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Learning Disorders; Executive Dysfunction
Keywords: Executive Functions; learning disorder; children
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: the study was carried on a single group underwent initial assessment then intervention then final assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): single group who had intervention and comparison of pre and post intervention assessment
  Interventions: Other: Executive functions training-elementary and Promoting executive function in in the classroom

INTERVENTIONS:
Other: Executive functions training-elementary and Promoting executive function in in the classroom — evidence based practice that target executive function skills in early elementary years.

SUMMARY:
In recent years, significant progress has been made on ways to improve Executive Functions (EF) skills for school readiness involving direct EF training and classroom educational programs. Due to the absence of a well-structured Arabic program for EF training in children, the rationale of this study is to implement a comprehensive, evidence-based intervention program to help Egyptian children with learning disorders to overcome their EF impairment. It uses the multimodality approach to help meet the needs of students with a variety of learning styles. The aim of this study is to adapt the combined form of the "Executive Functions Training-Elementary", and the "Promoting Executive Function In The Classroom" programs and its application in order to test its effectiveness in the rehabilitation of Egyptian learning disordered children.

DETAILED DESCRIPTION:
The study was conducted on 40 children with dyslexia and Executive dysfunction attending unit of phoniatrics, Otorhinolaryngology department, Alexandria University. The results were compared before and after intervention.

The "Executive Functions Training-Elementary" program is an evidence-based practice that targets Executive function skills in the early elementary years by training students how to plan, execute, complete, and monitor tasks. It develops cognitive abilities and behavior control with classroom-related activities for varying ability levels.

The "Promoting Executive Function In The Classroom" program helps to incorporate Executive function processes (such as planning, organization, prioritizing, and self-checking) into the classroom curriculum. Chapters provide effective strategies for learning by improving how to learn.

Data were collected and entered to the computer using (Statistical Package for Social Science) program for statistical analysis (version 21).

Data were entered as numerical or categorical, as appropriate. Kolmogorov-Smirnov test of normality revealed no significance in the distribution of the variables, so the parametric statistics was adopted.

Data were described using minimum, maximum, mean, standard deviation and 95% Confidence Interval of the mean.

Categorical variables were described using frequency and percentage. Comparisons were carried out between two studied dependent normally distributed variables using paired t-test.

Comparisons were carried out between more than two independent normally distributed subgroups using one-way Analysis Of Variance (ANOVA) test. When F ratio of ANOVA was significant Levene test of homogeneity of variances was done, and if significant Brown-Forsythe Robust test was adopted. Post-hoc multiple comparisons was done using Games-Howell.

ELIGIBILITY:
Inclusion Criteria:

* children complaining of specific learning disorder and executive function deficits

Exclusion Criteria:

* brain damage, mentally retarded or history of fits or subclinical fits
* hearing or visual impairment
* psychic problems

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Self-Management to Time. | 3-6 months
  scored from 1-4 depending on the parent's answers concerning the child's performance in this item in the last 6 months
Self-Organization and Problem-Solving | 3-6 months
  scored from 1-4 depending on the parent's answers concerning the child's performance in this item in the last 6 months
Self-Restraint. | 3-6 months
  scored from 1-4 depending on the parent's answers concerning the child's performance in this item in the last 6 months
Self-Motivation. | 3-6 months
  scored from 1-4 depending on the parent's answers concerning the child's performance in this item in the last 6 months
Self-Regulation of Emotion | 3-6 months
  scored from 1-4 depending on the parent's answers concerning the child's performance in this item in the last 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Reham M Elmaghraby, MD, Study Chair — otorhinolaryngology department, Faculty of Medicine, Alexandria University; Engy S Elhakeem, MD, Study Director — otorhinolaryngology department, Faculty of Medicine, Alexandria University; Soha AL Ibrahim, MD, Study Chair — Neuropsychiatry department, Faculty of Medicine, Alexandria University
Locations (1):
- Faculty of Medicine, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All statistical data are available in the study once published
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publishing
Access Criteria: through the email address engy.elhakeem@alexmed.edu.eg

REFERENCES:
- [Background] Barbosa T, Rodrigues CC, Mello CB, Silva MCSE, Bueno OFA. Executive functions in children with dyslexia. Arq Neuropsiquiatr. 2019 May 13;77(4):254-259. doi: 10.1590/0004-282X20190033. PMID 31090806
- [Background] 3. Medapati N, Periasamy A. Comparing efficiency of executive functions between players and non-players of organized sport. Int J Physiol Nutr Phys Educ 2019; 1: 75-8.
- [Background] Doebel S. Rethinking Executive Function and Its Development. Perspect Psychol Sci. 2020 Jul;15(4):942-956. doi: 10.1177/1745691620904771. Epub 2020 Apr 29. PMID 32348707
- [Background] Cortes Pascual A, Moyano Munoz N, Quilez Robres A. The Relationship Between Executive Functions and Academic Performance in Primary Education: Review and Meta-Analysis. Front Psychol. 2019 Jul 11;10:1582. doi: 10.3389/fpsyg.2019.01582. eCollection 2019. PMID 31354585
- [Background] Baddeley A. Working memory: theories, models, and controversies. Annu Rev Psychol. 2012;63:1-29. doi: 10.1146/annurev-psych-120710-100422. Epub 2011 Sep 27. PMID 21961947
- [Background] Nguyen T, Duncan G J. Kindergarten components of executive function and third grade achievement: A national study. Early Childhood Res Q 2018; 2:1-13
- [Background] Op den Kelder R, Van den Akker AL, Geurts HM, Lindauer RJL, Overbeek G. Executive functions in trauma-exposed youth: a meta-analysis. Eur J Psychotraumatol. 2018 May 3;9(1):1450595. doi: 10.1080/20008198.2018.1450595. PMID 33488998
- [Background] Alsaedi RH, Carrington S, Watters JJ. Behavioral and Neuropsychological Evaluation of Executive Functions in Children with Autism Spectrum Disorder in the Gulf Region. Brain Sci. 2020 Feb 22;10(2):120. doi: 10.3390/brainsci10020120. PMID 32098341
- [Background] Lensing N, Elsner B. Development of hot and cool executive functions in middle childhood: Three-year growth curves of decision making and working memory updating. J Exp Child Psychol. 2018 Sep;173:187-204. doi: 10.1016/j.jecp.2018.04.002. Epub 2018 May 7. PMID 29734050
- [Background] Sung J, Wickrama K. Longitudinal relationship between early academic achievement and executive function: Mediating role of approaches to learning. Contemp Educ Psychol 2018; 24: 171-83
- [Background] Duran C, Byers A, Cameron CE, Grissmer D. Unique and compensatory associations of executive functioning and visuomotor integration with mathematics performance in early elementary school. Early Child Res Q 2018; 42: 21-30.
- [Background] Huang Y, He M, Li A, Lin Y, Zhang X, Wu K. Personality, Behavior Characteristics, and Life Quality Impact of Children with Dyslexia. Int J Environ Res Public Health. 2020 Feb 22;17(4):1415. doi: 10.3390/ijerph17041415. PMID 32098297
- [Background] Hebert M, Kearns DM, Hayes JB, Bazis P, Cooper S. Why Children With Dyslexia Struggle With Writing and How to Help Them. Lang Speech Hear Serv Sch. 2018 Oct 24;49(4):843-863. doi: 10.1044/2018_LSHSS-DYSLC-18-0024. PMID 30458545
- [Background] Meixner JM, Warner GJ, Lensing N, Schiefele U. The relation between executive functions and reading comprehension in primary-school students: A cross-lagged-panel analysis. Early Childhood Res Q 2018; 46: 1-13.
- [Background] Cragg L, Keeble S, Richardson S, Roome HE, Gilmore C. Direct and indirect influences of executive functions on mathematics achievement. Cognition. 2017 May;162:12-26. doi: 10.1016/j.cognition.2017.01.014. Epub 2017 Feb 9. PMID 28189034
- [Background] Nesbitt KT, Fuhs MW, Farran DC. Stability and instability in the co-development of mathematics, executive function skills, and visual-motor integration from prekindergarten to first grade. Early Childhood Res Q 2018; 1:1-13.